CLINICAL TRIAL: NCT04026477
Title: Evaluation of Link for Equity: A Program to Reduce Racial/Ethnic School Violence Disparities (School Staff Population)
Brief Title: Evaluation of Link for Equity (School Staff Population)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00007052; 1R01MD013801-01 (NIH)
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Universal Trauma-Informed Care and Cultural Humility Training (Experimental): Universal Trauma-Informed Care and Cultural Humility Training. After video and workshop training, staff will have ability to recognize trauma and racism and its impact on school procedures, practices, and children themselves. Staff will be able to apply core principles of cultural humility. Staff will examine their own cultural identity and how it influences their interactions and relationships with students of diverse cultural backgrounds (Principle 1). Staff will learn ways that privilege and oppression relate to their cultural identity and identify ways to flatten power hierarchies between themselves and students, including handling misbehavior from a trauma-informed, culturally humble perspective (Principle 2). Staff will problem-solve ways for their schools to be accountable for equitable discipline practices (Principle 3).
  Interventions: Behavioral: Immediate Universal Trauma-Informed Care and Cultural Humility Training
- Waitlist Universal Trauma-Informed Care and Cultural Humility Training (Active Comparator): All staff from waitlisted schools will receive Universal Trauma-Informed Care and Cultural Humility Training at the end of the waitlist period.
  Interventions: Behavioral: Waitlisted Universal Trauma-Informed Care and Cultural Humility Training

INTERVENTIONS:
Behavioral: Immediate Universal Trauma-Informed Care and Cultural Humility Training — Instructional video and workshop
  Arms: Immediate Universal Trauma-Informed Care and Cultural Humility Training
Behavioral: Waitlisted Universal Trauma-Informed Care and Cultural Humility Training — Instructional video and workshop following waitlist period
  Arms: Waitlist Universal Trauma-Informed Care and Cultural Humility Training

SUMMARY:
The investigators propose to develop and evaluate Link for Equity, a trauma-informed system of care. Link, a system of support for ACE-affected children, is composed of universal school Trauma-Informed Care. Preventing Racism through Awareness and Action (PRAA) is a perspective-taking racism/discrimination prevention intervention for school staff that increases awareness of racism and how it impacts students and promotes empathy for students of color. Link for Equity will be translated to be culturally responsive for 12 secondary public schools in metropolitan and rural Minnesota with substantial racial/ethnic minority students and racial/ethnic disparities in school discipline and violence. Using a nested, rigorous, and ethically acceptable randomized waitlist control design, the investigators will implement and evaluate Link for Equity sequentially for two years in each school. The overall goal is to evaluate if Link for Equity can reduce school violence disparities.

DETAILED DESCRIPTION:
Significance of Research Question/Purpose: Youth violence is an emergent nationwide public health issue. Almost two-thirds of public schools across America report one or more violent incidents on their campus annually. In 2014, approximately 850,000 non-fatal victimizations occurred among 12-18 year-old students; this includes 486,400 assaults and serious violent victimizations. About 22% of children in the U.S. reported being bullied at school in 2011, and one in 10 students report being threatened or injured with a weapon on school property in the past year.

Racial/ethnic minority youth are at increased risk for school violence. African American, Latino, and American Indian youth report higher rates of in-school physical fighting, weapon carrying, and gang presence compared to white youth. The highest rates of severe violence are reported in urban high schools with high minority enrollment, and large samples and reviews indicate Black and Latino youth engage in more bullying than other racial groups.

Accumulation of adverse child experiences (ACEs), or childhood traumas such as abuse, neglect, household dysfunction, and racial discrimination, place children at high risk for violent behaviors. Multiple ACEs are more prevalent among American Indian (40%), Hispanic (31%) and black children (33%) compared with white children (21%). ACEs have acute and cumulative detrimental impacts on the physiological, cognitive, behavioral and psychological health of children, and children with increased ACEs are more likely to engage in violent behaviors at school.

For example, the Olweus Anti-bullying Program, which was shown to be effective in Norway yet ineffective among Washington's racial/ethnic minority students, is implemented widely. A number of gaps in addressing risks for youth violence remain. Many programs are limited to didactic instruction in the classroom, or solely target children with significant behavioral concerns. Systems-based approaches are the most promising sustainable models because they capitalize on infrastructures and services offered at school. This study will evaluate a systems-based model, Link for Equity. Link is combines Trauma-Informed Care (TIC) and psychological first aid in a culturally sensitive manner. Link for Equity offers cultural humility training that specifically targets racial/ethnic microaggressions to prevent racial discrimination in discipline referrals of racial and ethnic minority students.

The aims are to:

Aim 1: Adapt, implement, and measure the effect of Link for Equity on school violence disparities.

Aim 2: Measure the effect of Link for Equity on racial discrimination by teachers (2a), and assess if teachers' racial discrimination mediates the effect of Link for Equity on school violence (2b).

Aim 3: Explore connectedness and stress mechanisms through which Link for Equity impacts school violence disparities.

ELIGIBILITY:
Inclusion Criteria:

* Employees of the participating school districts
* Willingness to complete study surveys

Exclusion Criteria:

* School staff not employees of the participating school districts
* School staff who refuse to complete study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1612 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Change in Color Blind Racial Attitudes Scale (CoBRAS) Score | baseline and 2 years
  This is a 20-item scale that measures denial of racism and white privilege and rejection of the belief that action is needed to eradicate the negative consequences of racism. Items are scored on a scale from 1 (strongly disagree) to 6 (strongly agree). Total scores are calculated by summing scores from all 20 items. Possible total scores range from 20-120 with higher scores indicating a stronger attitude of color-blindness.
Change in Acceptability of Racial Microaggressions Scale (ARMS) Score | baseline and 2 years
  Attitudes towards racial microaggressions will be measured using two subscales of the Acceptability of Racial Microaggressions Scale (ARMS): Color Evasion and Power Evasion. The Color Evasion subscale contains 8 statements and the power evasion subscale contains 7 statements, which staff score for appropriateness on a scale of 1 to 6. The scores for the Color Evasion subscale are averaged. The resulting score ranges from 1 to 6, with a higher score indicating higher acceptability of color evasion microaggressions. Likewise, the Power Evasion subscale scores are average, with final scores ranging from 1 to 6, and higher scores indicating a higher acceptability of power evasion microaggressions.
Change in Attitudes Related to Trauma-Informed Care Scale (ARTIC) Score | baseline and 2 years
  Attitudes related to trauma-informed care will be measured with the Attitudes Related to Trauma-Informed Care Scale (ARTIC), developed by the Traumatic Stress Institute. The ARTIC-10 Education version is a validated measure containing 10 questions answered on a bipolar Likert scale from 1 to 7. Certain items are reversed, and the item scores are averaged. Final scores range from 1 to 7, with higher scores indicating more favorable attitudes related to trauma-informed care.
Change in Scale of Ethnocultural Empathy Score | baseline and 2 years
  Ethnocultural Empathy will be measured using the validated Scale of Ethnocultural Empathy. The scale contains 31 statements, rated from 1 (strongly agree that this describes me) to 6 (that strongly disagree that this describes me). Certain items are reversed, and the item scores are averaged. Final scores range from 1 to 6, with higher scores indicating higher levels of ethnocultural empathy.

CONTACTS AND LOCATIONS:
Overall Officials: Marizen Ramirez, PhD, MPH, Principal Investigator — University of Minnesota; Andrew Ryan, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez MR, Ryan A, Harding AB, Renfro T, Church TR, Rosebush C, Trotter AG, Xiong BN, Gonzalez J, Woods-Jaeger B. Link for Equity, a community-engaged waitlist randomized controlled trial of a culturally responsive trauma-informed care program for BIPOC students: Design features and characteristics of baseline sample. Contemp Clin Trials. 2023 Mar;126:107090. doi: 10.1016/j.cct.2023.107090. Epub 2023 Jan 18. PMID 36681238